CLINICAL TRIAL: NCT01965691
Title: Application of Stable Isotopes to Determine Protein Requirements in Children With Phenylketonuria (PKU)
Brief Title: Protein Requirements in Children With Phenylketonuria (PKU)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Rare Disease Foundation, Vancouver, Canada (Other); Saudi Arabian Cultural Bureau, Ottawa (Unknown)
Responsible Party: Principal Investigator, Rajavel Elango, PhD, Principle Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: H13-00220
Record Dates: First submitted 2013-10-16; First posted 2013-10-18 (Estimated); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Phenylketonuria
Keywords: Phenylketonuria; PKU; Phenylalanine metabolism; Protein requirements; Indicator Amino acid Oxidation; Stable isotopes
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Protein intake (Experimental): Protein intake- Dietary supplement
  Interventions: Dietary Supplement: Protein intake

INTERVENTIONS:
Dietary Supplement: Protein intake — Oral consumption of eight hourly experimental meals-
  * 4 tracer free experimental meals containing a mixture of free amino acids and calories from protein free flavored liquid, protein free cookies and corn oil
  * 4 isotopically labeled experimental meals.

SUMMARY:
Phenylketonuria (PKU) is an inherited inborn error of an amino acid phenylalanine (PHE) metabolism affecting 1:15,000 births. It is caused by a decreased activity of an enzyme in the liver called phenylalanine hydroxylase (PAH) which is important to convert PHE into tyrosine, another amino acid. Consequently, PHE accumulates in the blood leading to mental and developmental delays. Nutritional management is the primary choice of treatment that includes providing sufficient protein in the diet and at the same time restricting PHE. However the amount of protein to be given is unknown. A new technique called Indicator Amino Acid Oxidation (IAAO) will be used to determine the protein requirements in children with PKU (5-18y). The study will help treat and manage these children with sufficient protein to ensure proper growth and development. Current dietary recommendations range from 35-65 g/day and is based on factorial calculations.

The investigators hypothesize that the protein requirement in children with PKU will be higher than the current mathematically calculated recommended intake of 35-65 g/day for the 5-18y children.

ELIGIBILITY:
Inclusion Criteria:

* Children (5-18y) who are diagnosed with Phenylketonuria (PKU), and clinically stable with no acute illness

Exclusion Criteria:

* Children less than 5y of age and who are diagnosed with PKU, as it may be difficult to take breath samples and perform indirect calorimetry in very young children.
* Children diagnosed with PKU, but are currently ill, with a fever, cold, vomiting or diarrhea.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2013-10; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
13 Co2 production | 8 hours (1 study day)
  Urine and breath samples will be collected during the study to measure the rate of oxidation of tracer in the expired breath and flux enrichment in urine.

CONTACTS AND LOCATIONS:
Overall Officials: Rajavel Elango, PhD, Principal Investigator — Child and Family Research Institute, University of British Columbia; Sylvia Stockler-Ipsiroglu, MD, Study Chair — University of British Columbia; Keiko Ueda, MPH, RD, Study Chair — Provincial Health Services Authority British Columbia
Locations (1):
- Child and Family Research Institute, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Turki A, Ueda K, Cheng B, Giezen A, Salvarinova R, Stockler-Ipsiroglu S, Elango R. The Indicator Amino Acid Oxidation Method with the Use of l-[1-13C]Leucine Suggests a Higher than Currently Recommended Protein Requirement in Children with Phenylketonuria. J Nutr. 2017 Feb;147(2):211-217. doi: 10.3945/jn.116.240218. Epub 2017 Jan 4. PMID 28053173